CLINICAL TRIAL: NCT07150598
Title: Immune-Marker Platform for Patients With Advanced Lung Cancer
Acronym: IMPALUX
Status: Not yet recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Wermke, Prof. Dr. med., Technische Universität Dresden
Other Study IDs: BO ff (Multi)-EK-118032025; DRKS00037281 (Other: German Clinical Trials Register (DRKS))
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); NSCLC Stage IIIB~IV; NSCLC Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Immunochemotherapy; Multiplex Immunofluorescence; 3'-RNA Sequencing; Prospective Observational Study; Tumor Microenvironment; Therapy Response; Precision Oncology
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will retain tumor biopsy specimens from patients with advanced non-small cell lung cancer (NSCLC). The samples include:
  Formalin-fixed, paraffin-embedded (FFPE) tumor tissue blocks or slides suitable for multiplex immunofluorescence staining and 3'-RNA sequencing analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kohort A: Patients with advanced non-small cell lung cancer (NSCLC) who undergo tumor biopsy at initial diagnosis and a second biopsy approximately 6 weeks after starting standard-of-care immunochemotherapy. Biospecimens will be analyzed using multiplex immunofluorescence and 3'-RNA sequencing to study immune and tumor-associated biomarkers.
- Kohort B: Patients with advanced NSCLC who undergo tumor biopsy at the time of disease progression or therapy line change while receiving standard-of-care immunochemotherapy. Biospecimens will be analyzed using multiplex immunofluorescence and 3'-RNA sequencing to study immune and tumor-associated biomarkers.

SUMMARY:
The goal of this observational study is to better understand how the immune system and certain tumor markers are linked to treatment response in patients with advanced non-small cell lung cancer (NSCLC) who receive immunochemotherapy.

The investigators aim to answer the following questions:

* Can the investigators successfully analyze immune markers and gene activity from small tumor samples (biopsies)?
* Are these markers connected to how well patients respond to immunochemotherapy and how their disease progresses?

What will participants do?

* Provide tumor tissue samples (biopsies) at key points: before treatment, about 6 weeks after starting immunochemotherapy, and if the cancer grows or treatment changes.
* Allow their tumor samples to be analyzed in the lab using advanced techniques to measure immune and genetic markers.
* Share clinical information (such as treatment response and disease progression) so investigators can study how it relates to these markers.

This study does not test a new drug or treatment.

ELIGIBILITY:
Inclusion Criteria:

For all:

* Written informed consent of the patient
* Consent of participation in the national Network for Genomic Medicine in Lung Cancer (nNGM)
* Advanced lung cancer with non-curative treatment option (NSCLC)
* No targetable driver mutation detected, defined as no targetable drive mutation in ALK, EGFR, BRAF, HER2, MET, NTRK, RET, ROS1
* PD-L1 expression on tumor cells (TPS < 50%)

Cohort A:

* Previously untreated NSCLC without curative treatment options
* Sufficient pre-treatment tumor material available for the planned analyses or consenting and able to undergo additional pretreatment biopsy
* Scheduled to undergo immune(chemo)therapy
* Willing and able to undergo re-biopsy 6 weeks after start of immune(chemo)therapy

Cohort B:

* Any line of progression after firstline immune(chemo)therapy
* Sufficient tumor material obtained after progression on most recent line of treatment available or willing and able to undergo re-biopsy prior to next line treatment

Exclusion Criteria:

* Any condition representing an unjustified risk for obtaining an additional biopsy sample (if needed) in the view of the investigator
* Incapability of understanding the purpose and possible consequences of the trial
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's cooperation with the requirements of the trial or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult patients (≥18 years) with histologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC) who are initiating or receiving standard-of-care immunochemotherapy. Eligible participants must be able to provide tumor biopsy material at predefined time points (baseline, 6 weeks after treatment start, and/or at progression or therapy line change). Both male and female patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
General technical success rate for multiplex immunofluorescence staining per biopsy | From enrollment until completion of all planned biopsy time points (baseline, 6 weeks after start of immunochemotherapy, and at each progression or therapy line change), up to approximately 24 months.
  defined as a staining, which is:
  1. considered evaluable by a trained pathologist according to the HE-, and multiplex-stained overview
  2. PanCK positive
  3. for which negative control and positive control stained in the same run are negative and positive, respectively.
  Estimated at 60 %.
General success rate for the 3'RNA-Sequencing Approach per biopsy | From enrollment until completion of all planned biopsy time points (baseline, 6 weeks after start of immunochemotherapy, and at each progression or therapy line change), up to approximately 24 months.
  defined as
  1. successful 3'RNA-isolation and -sequencing,
  2. keratin 18 (KRT18) expression is clearly detected above background, e.g. above a 5 Counts per million (CPM) cutoff and
  3. is considered evaluable by trained molecular biologist according to the sequencing results.
  For 3'RNA-Seq, gene-specific expression distributions will be used to calibrate CPM, ranks, or similar metric cutoffs to define positivity/negativity.
  Estimated at 60 %.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wermke, Prof. Dr., Principal Investigator — Medizinische Klinik I, Universitätsklinikum Carl Gustav Carus, Dresden; Jürgen Wolf, Prof. Dr., Principal Investigator — Klinik I für Innere Medizin, CIO, Universitätsklinikum Köln
Locations (2):
- Germany (2):
  - Universitätsklinikum Köln, Centrum für Integrierte Onkologie (CIO) Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No